CLINICAL TRIAL: NCT06128109
Title: An Exploratory, Prospective, Randomized, Subject and Evaluator-blinded, Split-face, Single-centre Trial Investigating the Effectiveness and Safety of THIODERM STRONG Compared to Juvéderm® VOLUMA® Lidocaine for the Treatment of Midface Volume Deficit (TIMI)
Brief Title: THIODERM STRONG Compared to Juvéderm® VOLUMA® Lidocaine for the Treatment of Midface Volume Deficit
Acronym: TIMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Collaborators: Proinnovera GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPH-50501
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Mid Face Volume Deficit
Keywords: Midface; Volume Deficit; Hyaluronic Acid; Dermal Filler

STUDY DESIGN:
Intervention Model Description: Split-Face Design with random assignment of test device and comparator device to be injected either into right or into left Mid Face Area
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and Evaluating Investigator will be blinded to study device assignment. The subject will be blind-folded during treatment. The Evaluating Investigator is unaware of the device assignment and has no access to study data that could potentially contain unblinding information
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group THIODERM LEFT (Other): Split Face Design: Test Device left midface and Comparator Device right midface
  Interventions: Device: Thioderm Strong; Device: Juvéderm VOLUMA Lidocaine
- Group JUVÈDERM LEFT (Other): Split Face Design: Test Device right midface and Comparator Device left midface
  Interventions: Device: Thioderm Strong; Device: Juvéderm VOLUMA Lidocaine

INTERVENTIONS:
Device: Thioderm Strong — Test Device
Device: Juvéderm VOLUMA Lidocaine — Comparator Device

SUMMARY:
This mono-center clinical investigation is intended to evaluate the safety and effectiveness of THIODERM STRONG (test device) in the correction of moderate to severe midface volume deficit compared to Juvéderm® VOLUMA® Lidocaine (comparator device).

DETAILED DESCRIPTION:
The Investigation is an exploratory, prospective, randomized, subject and evaluator-blinded, split- face, single-centre study investigating the effectiveness and safety of THIODERM STRONG compared to Juvéderm® VOLUMA® Lidocaine for the treatment of moderate to severe midface volume deficit. 20 eligible Subjects will be included in this investigation, after the informed consent form (ICF) has been signed and relevant pre-treatment procedures, including medical history and pregnancy testing, have been performed. Subjects will receive injection in the midface region using THIODERM STRONG and Juvéderm® VOLUMA® Lidocaine until an optimal aesthetic result is achieved. The Blinded Evaluating Investigator will determine severity of the Subject's midface volume deficit using the 5-point MVDSS throughout the investigation (Baseline to Week 24). Baseline is defined as the assessment prior to administration of the IMDs. The same Investigator will assess the Subject using the 5-point MVDSS at all visits. An optional touch-up treatment can be performed at Week 4 upon discretion of the Unblinded Treating Investigator. The effectiveness and safety of the treatment will be evaluated after Day 1, 3 and 7 as well as at 4, 8, 16 and 24 weeks using objective and subjective outcome parameters. An interim analysis will be performed when all Subjects have completed the visit at Week 8.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at the time of screening (upper limit 75 years, inclusive).
2. Subjects with bilateral, approximately symmetric moderate to severe midface volume deficit (severity scores of 2 or 3 on the 5-point Midface Volume Deficit Severity Scale), shown by the same rating on both sides, assessed by the Blinded Evaluating Investigator.
3. Healthy skin in the midface area and free of diseases that could interfere in cutaneous aging evaluation.
4. Subject has a stable medical condition with no uncontrolled systemic disease.
5. Females of childbearing potential must have a negative urine pregnancy test and must agree to use a highly effective method of birth control throughout the entire study1.
6. Male subjects with female partners of child-bearing potential must agree to use contraception throughout the entire study (surgical sterilization or a physical barrier such as a condom).
7. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of study, including botulinum toxin injection (except glabella or forehead botulinum toxin treatment).
8. Subjects who understand the purpose and conduct of the study and having given written informed consent and are willing and able to attend the study visits as judged by the Investigator.

Exclusion Criteria:

1. Females, who are pregnant and/or, lactating or planning to become pregnant during the clinical investigation.
2. History of allergies or hypersensitivity to hyaluronic acid and/or to gram positive bacterial proteins, lidocaine, or any amide-based anaesthetic
3. History of severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies.
4. Tendency to keloid formation and/or hypertrophic scars.
5. Presence of infectious, inflammatory, or proliferative cancerous or pre-cancerous lesions in the area to be treated.
6. Recurrent (three times a year over the last year) herpes simplex in the treatment areas
7. Known human immune deficiency virus-positive individuals.
8. History or presence of any autoimmune or connective tissue disease
9. Uncontrolled (or unstable) Diabetes mellitus or uncontrolled systemic diseases as per Investigator discretion.
10. Previous facial plastic surgery, tissue augmentation with silicone, fat or another non-absorbable substance (permanent fillers) and semi-permanent / long-lasting fillers (e.g., poly-L-lactic acid (PLLA), Polymethylmethacrylate (PMMA) filler) in the area of device application and during the entire investigation
11. Implantation of dermal fillers in the treatment area within the preceding 24 months prior to Visit 0 (Screening) and during the entire investigation
12. Subject has received any of the following aesthetic treatments in the midface area: e.g., laser therapy, absorbable and non-absorbable sutures (threads), dermabrasion, mesotherapy, micro-needling and/or botulinum toxin (including treatment of crow´s feet in the outer eye region) within the last 12 months prior to Visit 1, chemical peeling within the last three months prior to Visit 1 or is planning to undergo such procedures during entire investigation
13. Facial lipolysis, including submental fat treatments, within the previous 12 months prior to Visit 0 (Screening) and during the entire investigation
14. Bariatric surgery within 12 months prior to Visit 0 (Screening) and during the entire investigation.
15. History of bleeding disorder and/or use of anticoagulant, antiplatelet or thrombolytic medication, including nutrition supplements that potentially prolong coagulation, from 10 days pre- to 3 days post-injection (initial treatment and touch-up treatment).
16. Systemic glucocorticoids, including immunosuppressant or immunomodulators, within 8 weeks prior to undergoing investigational device injections.
17. Patients suffering from untreated epilepsy.
18. Patients with acute rheumatic fever with heart complications.
19. Patients with symptoms of cardiac conduction disorders.
20. Planned dental/oral surgery or modification (bridgework, implants) within four weeks prior to each injection and to a minimum of four weeks post injection (initial treatment, touch-up treatment).
21. Beard longer than three-day beard, or excessive facial hair that could interfere in evaluation of treatment as judged by the Investigator.
22. Subjects with active SARS-CoV-2019 infection and Subjects with symptoms consistent with COVID-19 infection including any other respiratory symptoms/illnesses within the past 14 days unless tested negative prior to Visit 0 (Screening).
23. Any medical condition prohibiting the inclusion in the clinical investigation according to the judgment of the Investigator.
24. Previous enrolment in this clinical investigation.
25. Current participation in another clinical investigation, or treatment with any investigational drug/medical device within 30 days prior to clinical investigation Visit 0 (Screening), or 5 half-lives of the investigational drug, whichever is longer.
26. Midface volume deficit due to a congenital defect, trauma, or abnormalities in facial adipose tissue distribution such as those associated with HIV related lipodystrophy.
27. Subjects who experienced fat loss for a minimum of 10% of body weight over the last 12 months (e.g., post bariatric patients), or Subjects who have the intention to change eating habits that result in a weight gain or loss >10% during the entire investigation.
28. Close affiliation with the Investigator (e.g., a close relative, financially dependent on the study site) or Subject who is an employee of the Sponsor's company or group companies of the Sponsor.
29. Any individual whose willingness to volunteer in this clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Response Magnitude | 24 Weeks
  To assess the effectiveness of THIODERM STRONG in reducing the severity of the midface volume deficit in comparison with Juvéderm® VOLUMA® Lidocaine based on Blinded Evaluating Investigator assessment at Week 24 as measured via the 5-point Midface Volume Deficit Severity Scale (MVDSS).

SECONDARY OUTCOMES:
Total Volume Injected | 24 Weeks
  To assess required total volume for optimum aesthetic result for THIODERM STRONG compared to Juvéderm® VOLUMA® Lidocaine.
Response Rate | Day7; Week 4, 8, 16, and 24
  To assess the proportion of responders after treatment with THIODERM STRONG in comparison with Juvéderm® VOLUMA® Lidocaine per treated side.
Response Magnitude | Day 7; Week 4, 8, and 16
  To assess the change on the 5-point MVDSS from baseline after treatment with THIODERM STRONG in comparison with Juvéderm® VOLUMA® Lidocaine.
Response Magnitude Photographic Review | Day7; Week 4, 8, 16, and 24
  Change of 5-point MVDSS from baseline to Day 7 and Week 4, 8, 16 and 24 based on the independent blinded evaluating panel's assessment per treated side.
Aesthetic Improvement via GAIS - Investigator | Day7; Week 4, 8, 16, and 24
  Aesthetic improvement based on the Blinded Evaluating Investigator's assessment per treated side at Week 4, 8, 16 and 24 using the GAIS.
Aesthetic Improvement via GAIS - Subject | Day7; Week 4, 8, 16, and 24
  Aesthetic improvement based on the Subject's assessment per treated side at Week 4, 8, 16 and 24 using the GAIS
Volume Change via 3D Imaging | Day7; Week 4, 8, 16, and 24
  Volume change of the midface region at Day 7 and Week 4, 8, 16 and 24, based on 3D surface imaging in comparison to the baseline 3D surface image per treated side.
Subject Satisfaction - Face-Q(TM) Outcome Scale | Day 1, 3, and 7; Week 4, 8, 16, and 24
  The extent of Subject´s satisfaction with treatment of the midface at Day 1, 3, 7 and Week 4, 8, 16 and 24 as assessed by the FACE-QTM Satisfaction with Outcome Scale per treated side.
Subject Appearance Appraisal - Face-Q(TM) Satisfaction with Cheeks | Day 1, 3, and 7; Week 4, 8, 16, and 24
  The extent of Subject´s appearance appraisal at Day 1, 3, 7 and Week 4, 8, 16 and 24 as assessed by the FACE-QTM Satisfaction with Cheeks Scale per treated side and compared to the score at screening.
Change of Nasolabial Fold Severity | Day7; Week 4, 8, 16, and 24
  Change of nasolabial fold severity measured by NLF-SRS from baseline to Day 7 and Week 4, 8, 16 and 24 based on the Blinded Evaluating Investigator's assessment per treated side.
Pain Assessment | Day 0; Week 4 (in case of touch-up treatment)
  Subject´s pain assessment after each treatment on an 11-point scale, where 0 is no pain and 10 is the worst pain imaginable per treated side.

OTHER OUTCOMES:
Safety Evaluation | through study completion, an average of 24 weeks
  Frequency, severity and causal relationship of adverse events (AEs) and serious adverse events (SAEs) during the entire study period, including adverse device effects (ADEs) and serious adverse device effects (SADEs).

CONTACTS AND LOCATIONS:
Overall Officials: Alice Krames-Juerss, Study Director — CROMA Pharma GmbH (Sponsor)
Locations (1):
- H&P Ambulatorien GmbH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No